CLINICAL TRIAL: NCT06211569
Title: Study of the Prevalence of Endometriosis and Adenomyosis in Women of Childbearing Age Consulting for Non-medical Oocyte Self-preservation
Brief Title: Study of the Prevalence of Endometriosis and Adenomyosis
Acronym: PrevADEOSE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231461; 2023-A01474-41 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Elective Fertility Preservation
Keywords: Endometriosis; Adenomyosis; Prevalence; Elective fertility preservation; Transvaginal pelvic ultrasound
MeSH Terms: conditions — Endometriosis; Adenomyosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Women of childbearing age, consulting for elective fertility preservation
  Interventions: Other: Usual follow-up

INTERVENTIONS:
Other: Usual follow-up — Usual follow-up

SUMMARY:
Our study aims to assess the prevalence of adenomyosis and endometriosis in patients consulting for elective fertility preservation through the diagnosis of these pathologies by transvaginal pelvic ultrasound. Imaging data will be compared with clinical data (patient characteristics, clinical symptoms) as well as the assessment of anxiety, depression, and quality of life collected from the women.

DETAILED DESCRIPTION:
Adenomyosis and endometriosis are two heterogeneous benign gynecological pathologies, in terms of the presence of diverse phenotypes and their symptomatic presentation: While some women are entirely asymptomatic, others experience pelvic pain, infertility, or abnormal uterine bleeding.

Assessing the prevalence of these two pathologies is challenging: On the one hand, a significant number of women are asymptomatic and not considered in the calculation; on the other hand, endometriosis and adenomyosis are often underdiagnosed, leading to delayed diagnosis.

Endometriosis and adenomyosis are frequently associated. Improving knowledge about the epidemiology of endometriosis and adenomyosis is crucial as both are major causes of clinical symptoms that adversely affect the quality of life in numerous women. This is a significant issue for women's health due to the associated suffering, numerous surgical interventions, healthcare expenses, and the suggested link with pathologies that may affect other organs. Understanding the disease could lead to improved treatment and the development of preventive strategies.

Therefore, it is urgent to determine the frequency of endometriosis and adenomyosis, as well as the correlation between women's characteristics, especially their clinical symptoms, and different phenotypes. In order to assess the prevalence of adenomyosis and endometriosis in a population of women of reproductive age, the investigators intend to conduct this single-center study focusing on patients consulting for non-medical fertility preservation.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged between 29 and 37
* Consultant for non-medical fertility preservation in the Reproductive Medicine Unit Port Royal, Cochin
* Informed and not opposed to this research
* Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant women
* Refusing to take part in the study
* Under court protection, curatorship or guardianship
* Women with a known malformation of the genital tract

Ages: 29 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women of childbearing age, not pregnant, consulting for non-medical oocyte self-preservation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Transvaginal pelvic ultrasound | Up to month 6
  Search for endometriosis and adenomyosis on transvaginal pelvic ultrasound and characterisation of lesions.

SECONDARY OUTCOMES:
Self-questionnaire | Inclusion
  Socio-demographic data
Self-questionnaire | Inclusion
  Medical history
Quality of life assessment (WHO-QOL-BREF) | Inclusion
  Between 26 (Poor quality of life) and 130 (good quality of life)
Hospital Anxiety and Depression Scale (HADS) | Inclusion
  2 scores between 0 (No anxiety or depression) and 21 (lots of anxiety and depression)

CONTACTS AND LOCATIONS:
Locations (1):
- Gynécologie Obstétrique II et médecine de la reproduction, Hôpital Cochin, Port Royal, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bird CC, McElin TW, Manalo-Estrella P. The elusive adenomyosis of the uterus--revisited. Am J Obstet Gynecol. 1972 Mar;112(5):583-93. doi: 10.1016/0002-9378(72)90781-8. No abstract available. PMID 5059589
- [Background] Bordonne C, Puntonet J, Maitrot-Mantelet L, Bourdon M, Marcellin L, Dion E, Plu-Bureau G, Santulli P, Chapron C. Imaging for evaluation of endometriosis and adenomyosis. Minerva Obstet Gynecol. 2021 Jun;73(3):290-303. doi: 10.23736/S2724-606X.21.04710-9. PMID 34008384
- [Background] Bourdon M, Oliveira J, Marcellin L, Santulli P, Bordonne C, Maitrot Mantelet L, Millischer AE, Plu Bureau G, Chapron C. Adenomyosis of the inner and outer myometrium are associated with different clinical profiles. Hum Reprod. 2021 Jan 25;36(2):349-357. doi: 10.1093/humrep/deaa307. PMID 33491057
- [Background] Bourdon M, Santulli P, Marcellin L, Maignien C, Maitrot-Mantelet L, Bordonne C, Plu Bureau G, Chapron C. Adenomyosis: An update regarding its diagnosis and clinical features. J Gynecol Obstet Hum Reprod. 2021 Dec;50(10):102228. doi: 10.1016/j.jogoh.2021.102228. Epub 2021 Sep 11. PMID 34520877
- [Background] Bulun SE. Endometriosis. N Engl J Med. 2009 Jan 15;360(3):268-79. doi: 10.1056/NEJMra0804690. No abstract available. PMID 19144942
- [Background] Chapron C, Marcellin L, Borghese B, Santulli P. Rethinking mechanisms, diagnosis and management of endometriosis. Nat Rev Endocrinol. 2019 Nov;15(11):666-682. doi: 10.1038/s41574-019-0245-z. Epub 2019 Sep 5. PMID 31488888
- [Background] Chapron C, Tosti C, Marcellin L, Bourdon M, Lafay-Pillet MC, Millischer AE, Streuli I, Borghese B, Petraglia F, Santulli P. Relationship between the magnetic resonance imaging appearance of adenomyosis and endometriosis phenotypes. Hum Reprod. 2017 Jul 1;32(7):1393-1401. doi: 10.1093/humrep/dex088. PMID 28510724
- [Background] Chapron C, Vannuccini S, Santulli P, Abrao MS, Carmona F, Fraser IS, Gordts S, Guo SW, Just PA, Noel JC, Pistofidis G, Van den Bosch T, Petraglia F. Diagnosing adenomyosis: an integrated clinical and imaging approach. Hum Reprod Update. 2020 Apr 15;26(3):392-411. doi: 10.1093/humupd/dmz049. PMID 32097456
- [Background] Di Donato N, Montanari G, Benfenati A, Leonardi D, Bertoldo V, Monti G, Raimondo D, Seracchioli R. Prevalence of adenomyosis in women undergoing surgery for endometriosis. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:289-93. doi: 10.1016/j.ejogrb.2014.08.016. Epub 2014 Aug 15. PMID 25201608
- [Background] Schwartz JC. Incidence of listeriosis in Pennsylvania livestock. J Am Vet Med Assoc. 1967 Dec 1;151(11):1435-7. No abstract available. PMID 5624198
- [Background] Fauconnier A, Chapron C. Endometriosis and pelvic pain: epidemiological evidence of the relationship and implications. Hum Reprod Update. 2005 Nov-Dec;11(6):595-606. doi: 10.1093/humupd/dmi029. Epub 2005 Sep 19. PMID 16172113
- [Background] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453
- [Background] Endo T, Kaneshige M, Nakazato M, Ohmori M, Harii N, Onaya T. Thyroid transcription factor-1 activates the promoter activity of rat thyroid Na+/I- symporter gene. Mol Endocrinol. 1997 Oct;11(11):1747-55. doi: 10.1210/mend.11.11.0012. PMID 9328356
- [Background] Hudelist G, Fritzer N, Thomas A, Niehues C, Oppelt P, Haas D, Tammaa A, Salzer H. Diagnostic delay for endometriosis in Austria and Germany: causes and possible consequences. Hum Reprod. 2012 Dec;27(12):3412-6. doi: 10.1093/humrep/des316. Epub 2012 Sep 17. PMID 22990516
- [Background] Khan KN, Fujishita A, Koshiba A, Kuroboshi H, Mori T, Ogi H, Itoh K, Nakashima M, Kitawaki J. Biological differences between intrinsic and extrinsic adenomyosis with coexisting deep infiltrating endometriosis. Reprod Biomed Online. 2019 Aug;39(2):343-353. doi: 10.1016/j.rbmo.2019.03.210. Epub 2019 Mar 27. PMID 31160242
- [Background] Kunz G, Beil D, Huppert P, Noe M, Kissler S, Leyendecker G. Adenomyosis in endometriosis--prevalence and impact on fertility. Evidence from magnetic resonance imaging. Hum Reprod. 2005 Aug;20(8):2309-16. doi: 10.1093/humrep/dei021. Epub 2005 May 26. PMID 15919780
- [Background] Leyendecker G, Bilgicyildirim A, Inacker M, Stalf T, Huppert P, Mall G, Bottcher B, Wildt L. Adenomyosis and endometriosis. Re-visiting their association and further insights into the mechanisms of auto-traumatisation. An MRI study. Arch Gynecol Obstet. 2015 Apr;291(4):917-32. doi: 10.1007/s00404-014-3437-8. Epub 2014 Sep 21. PMID 25241270
- [Background] Moradi Y, Shams-Beyranvand M, Khateri S, Gharahjeh S, Tehrani S, Varse F, Tiyuri A, Najmi Z. A systematic review on the prevalence of endometriosis in women. Indian J Med Res. 2021 Mar;154(3):446-454. doi: 10.4103/ijmr.IJMR_817_18. PMID 35345070
- [Background] Morassutto C, Monasta L, Ricci G, Barbone F, Ronfani L. Incidence and Estimated Prevalence of Endometriosis and Adenomyosis in Northeast Italy: A Data Linkage Study. PLoS One. 2016 Apr 21;11(4):e0154227. doi: 10.1371/journal.pone.0154227. eCollection 2016. PMID 27101396
- [Background] Naftalin J, Hoo W, Pateman K, Mavrelos D, Holland T, Jurkovic D. How common is adenomyosis? A prospective study of prevalence using transvaginal ultrasound in a gynaecology clinic. Hum Reprod. 2012 Dec;27(12):3432-9. doi: 10.1093/humrep/des332. Epub 2012 Sep 20. PMID 23001775
- [Background] Pinzauti S, Lazzeri L, Tosti C, Centini G, Orlandini C, Luisi S, Zupi E, Exacoustos C, Petraglia F. Transvaginal sonographic features of diffuse adenomyosis in 18-30-year-old nulligravid women without endometriosis: association with symptoms. Ultrasound Obstet Gynecol. 2015 Dec;46(6):730-6. doi: 10.1002/uog.14834. PMID 25728241
- [Background] Shigesi N, Kvaskoff M, Kirtley S, Feng Q, Fang H, Knight JC, Missmer SA, Rahmioglu N, Zondervan KT, Becker CM. The association between endometriosis and autoimmune diseases: a systematic review and meta-analysis. Hum Reprod Update. 2019 Jul 1;25(4):486-503. doi: 10.1093/humupd/dmz014. PMID 31260048
- [Background] Van den Bosch T, Dueholm M, Leone FP, Valentin L, Rasmussen CK, Votino A, Van Schoubroeck D, Landolfo C, Installe AJ, Guerriero S, Exacoustos C, Gordts S, Benacerraf B, D'Hooghe T, De Moor B, Brolmann H, Goldstein S, Epstein E, Bourne T, Timmerman D. Terms, definitions and measurements to describe sonographic features of myometrium and uterine masses: a consensus opinion from the Morphological Uterus Sonographic Assessment (MUSA) group. Ultrasound Obstet Gynecol. 2015 Sep;46(3):284-98. doi: 10.1002/uog.14806. Epub 2015 Aug 10. PMID 25652685
- [Background] Vercellini P, Vigano P, Somigliana E, Daguati R, Abbiati A, Fedele L. Adenomyosis: epidemiological factors. Best Pract Res Clin Obstet Gynaecol. 2006 Aug;20(4):465-77. doi: 10.1016/j.bpobgyn.2006.01.017. Epub 2006 Mar 24. PMID 16563868
- [Background] Yu O, Schulze-Rath R, Grafton J, Hansen K, Scholes D, Reed SD. Adenomyosis incidence, prevalence and treatment: United States population-based study 2006-2015. Am J Obstet Gynecol. 2020 Jul;223(1):94.e1-94.e10. doi: 10.1016/j.ajog.2020.01.016. Epub 2020 Jan 15. PMID 31954156